CLINICAL TRIAL: NCT00784667
Title: Dual Inhibition of EGFR Signalling Using the Combination of Cetuximab (Erbitux) and Erlotinib (Tarceva) in Patients With Chemotherapy-refractory Colorectal Cancer
Brief Title: Dual Inhibition of EGFR Signalling Using the Combination of Cetuximab and Erlotinib
Acronym: Dux
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Austin Health (Other Government)
Collaborators: Ballarat Health Services (Other); Queen Elizabeth Hospital, Adelaide (Unknown); Royal North Shore Hospital (Other)
Responsible Party: Dr Niall Tebbutt, Austin Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2008/03282
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2008-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal neoplasm; Metastasis
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Cetuximab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cetuximab — 400mg/m2 intravenously week 1, then 250 mg/m2 weekly intravenously
  Other Names: Erbitux
Drug: Erlotinib — 100mg orally daily continuously
  Other Names: Tarceva

SUMMARY:
This is a clinical trial investigating the effectiveness and safety of the combination of the study drugs cetuximab and erlotinib in patients with advanced (metastatic) refractory colorectal (bowel) cancer. If bowel cancer has spread to other organs (metastatic colorectal cancer), it is usually incurable and life-expectancy without treatment is less then 6 months on average. Currently, chemotherapy has been shown to have a significant impact in advanced colorectal cancer in terms of maintenance of quality of life and extension of survival. However, ultimately tumours will develop resistance to chemotherapy. Treatment options and subsequent survival at that stage are very limited. Therefore, new therapeutic approaches are urgently needed.

It is common for colorectal cancer cells to contain growth receptors, like antennae, on their surface which regulate their growth. The drugs used in this trial have been shown to be effective in targeting one of these growth receptors; the epidermal growth factor receptor (EGFR). Cetuximab is an antibody (protein produced by the immune system involved in the defense of the body against infections) against EGFR. Cetuximab has been shown to improve the survival of patients with chemotherapy refractory advanced colorectal cancer. Erlotinib is a protein that prevents activation and hence signaling by EGFR. Erlotinib improves survival in patients with advanced lung cancer. Although, each of these drugs are known to be effective at inhibiting EGFR when they are given alone, at least in some cases, it is hoped that using two drugs that target the same receptor pathway in different ways will provide a more effective treatment.

50 patients from four hospitals in Australia will participate in this trial, with approximately 25 patients being enrolled at Austin Health. All participants will receive the same treatment.

Neither of the study drugs are chemotherapy, and hence it is expected that the treatment would be well tolerated. The most frequent side effect associated with EGFR inhibitors is skin rash. Other possible side effects are diarrhea and low magnesium levels.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Histological diagnosis of colorectal cancer
* Metastatic disease not amenable to resection
* Measurable disease as assessed by CT scan using RECIST criteria
* Received and failed fluoropyrimidine therapy, where failure is defined as radiological progression after therapy for metastatic disease, prior adjuvant therapy, or toxicity limiting further therapy
* Received and failed oxaliplatin therapy, where failure is defined as radiological progression after therapy for metastatic disease, prior adjuvant therapy ,or toxicity (including neuro-toxicity) limiting further therapy
* Received and failed irinotecan therapy, where failure is defined as radiological progression after therapy for metastatic disease or toxicity limiting further therapy
* ECOG PS 0-1
* Adequate bone marrow function with platelets > 100 X 109/l; neutrophils > 1.5 X 109/l
* Adequate renal function, with calculated creatinine clearance >40 ml/min (Cockcroft and Gault).
* Adequate hepatic function with serum total bilirubin < 1.25 X upper limit of normal range and ALT or AST<2.5xULN (<5xULN if liver metastases present)
* Life expectancy of at least 12 weeks
* No other concurrent uncontrolled medical conditions
* No other malignant disease apart from non-melanotic skin cancer or carcinoma in situ of the uterine cervix or any other cancer treated with curative intent >2 years previously without evidence of relapse
* Women and partners of women of childbearing potential must agree to use adequate contraception
* Written informed consent including consent for biomarker studies

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent or to complete the protocol
* Prior treatment with drugs targeting EGFR such as cetuximab, panitumumab or erlotinib
* Participation in any investigational drug study within the previous 4 weeks
* Patients with uncontrolled clinically significant cardiac disease, arrhythmias or angina pectoris
* Untreated CNS metastases
* Pregnancy or lactation
* k-ras mutant tumours now excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
To determine the response rate (RECIST criteria). Responses will be evaluated for the whole patient group and separately for k-ras wild-type and k-ras mutant tumours | 6 weekly

SECONDARY OUTCOMES:
Toxicity | Weekly
Progression free survival | 6 weekly
Overall survival | Weekly

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Royal North Shore Hospital, Sydney, New South Wales
  - Queen Elizabeth Hospital, Adelaide, South Australia
  - Ballarat Base Hospital, Ballarat, Victoria
  - Austin Health, Melbourne, Victoria